CLINICAL TRIAL: NCT00150592
Title: A Phase II Study to Assess the Safety, Tolerability and Efficacy of SPD503 Administered to Children and Adolescents Aged 6-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety, Tolerability and Efficacy of SPD503 in Treating ADHD in Children Aged 6-17
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD503-206
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SPD503 (Guanfacine HCl) (Experimental)
  Interventions: Drug: SPD503 (Guanfacine HCl)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503 (Guanfacine HCl)
  Arms: SPD503 (Guanfacine HCl)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of SPD503 compared to placebo on tasks of sustained attention in children and adolescents aged 6-17 diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a primary diagnosis of ADHD
* Minimum baseline visit ADHD-RS-IV score of 24 and a baseline CGI-S score =>4
* Male or non-pregnant female subject who agrees to comply with any applicable contraceptive requirements
* Subject weighs > 55 lbs and is not morbidly overweight

Exclusion Criteria:

* Subject has a comorbid psychiatric diagnosis (except ODD) with significant symptoms such as any severe comorbid Axis II disorders or severe Axis I disorders
* Subject has a history of seizure disorder
* Subject has any specific cardiac condition or family history of significant cardiac condition
* Subject is pregnant, lactating or within six month post-partum

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2005-05-12 (Actual); Primary Completion 2005-10-05 (Actual); Study Completion 2005-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Kollins SH, Lopez FA, Vince BD, Turnbow JM, Farrand K, Lyne A, Wigal SB, Roth T. Psychomotor functioning and alertness with guanfacine extended release in subjects with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2011 Apr;21(2):111-20. doi: 10.1089/cap.2010.0064. Epub 2011 Apr 10. PMID 21476931
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 182 subjects were enrolled. Four (4) subjects were terminated prior to receiving study medication. Thus, 178 were randomized and received study medication.
Groups:
- SPD503: Subjects received either 1, 2, or 3 mg once-daily of SPD503 (Guanfacine hydrochloride) for 6 weeks.
Period: Overall Study
Arm/Group | SPD503 | Placebo
Started | 121 | 57
Completed | 114 | 54
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 | Placebo | Total
Number analyzed (Participants) | 121 | 57 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 121 | 57 | 178
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (2.83) | 12.8 (2.77) | 12.6 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 13 | 54
  Male | 80 | 44 | 124
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 57 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Choice Reaction Time (CRT) at 6 Weeks
Description: Choice reaction time (CRT) is a computerized assessment that trains the subject in holding down a press-pad and releasing the press-pad in response to stimuli presented on the screen. The task requires the subject to react as soon as a yellow dot appears in one of five locations, and the subject must respond by lifting their hand from the press-pad. This is the reaction time (RT) and ranges from 100 to 5000 msec. Lower scores indicate better performance.
Time Frame: Baseline and 6 weeks
Population: Per protocol (PP) defined as all subjects who completed the study and were deemed to be protocol-compliant.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 80 | 35
msec | 20.7 (63.11) | 21.9 (64.04)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.844, ANCOVA

2. Secondary Outcome: Change From Baseline in Digital Symbol Substitution Task/Coding Test (DSST/Coding) Scores at 6 Weeks in Age Category 8-17 Years
Description: The Digital Symbol Substitution Task/Coding Test (DSST/Coding) assesses relative contributions of speed, memory, and visual scanning. Subjects are required to copy symbols that are paired with simple geometric shapes or numbers within a specific time. Scores range from 0-65 in age category 6-7 years and 0-199 in age category 8-17 years. Higher scores indicate better performance.
Time Frame: Baseline and 6 weeks
Population: PP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 77 | 34
Units on a scale | 18.3 (14.03) | 20.7 (17.18)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.274, ANCOVA; Mean reaction time (adjusted) for each randomized treatment group at endpoint

3. Secondary Outcome: Change From Baseline in DSST/Coding Scores at 6 Weeks in Age Category 6-7 Years
Description: as for outcome 2
Time Frame: Baseline and 6 weeks
Population: PP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 3 | 1
Units on a scale | 1.9 (1.95) | 9.7 (0)

4. Secondary Outcome: Change From Baseline in Spatial Working Memory (SWM) Scores at 6 Weeks
Description: The Spatial Working Memory (SWM) Test is a computerized assessment of working memory and strategy performance. The subject is required to find blue "tokens" in various displayed boxes and use the "tokens" to fill a column on the right side of the screen. Subjects can only find "tokens" in new boxes, therefore they must remember where previous "tokens" were found. SWM scores including number of between errors, number of within errors, and number of double errors range 0-800 and SWM strategy scores range 8-56. Lower scores indicate better performance.
Time Frame: Baseline and 6 weeks
Population: PP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 80 | 35
Units on a scale
  Between errors | -4.4 (7.42) | -3.2 (6.75)
  Within errors | 0.0 (1.11) | -0.1 (0.73)
  Double errors | -0.0 (0.69) | 0.1 (0.53)
  Strategy | -0.9 (2.74) | -0.1 (2.56)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Between errors; Test type: Superiority or Other; p = 0.307, ANCOVA
Statistical Analysis 2: Comparison: SPD503 vs Placebo; Within errors; Test type: Superiority or Other; p = 0.552, ANCOVA
Statistical Analysis 3: Comparison: SPD503 vs Placebo; Double errors; Test type: Superiority or Other; p = 0.917, ANCOVA
Statistical Analysis 4: Comparison: SPD503 vs Placebo; Strategy; Test type: Superiority or Other; p = 0.068, ANCOVA

5. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Total Score at 6 Weeks
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set (FAS) defined as all subjects who received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 121 | 57
Units on a Scale | -8.8 (5.98) | -5.5 (7.23)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA

6. Secondary Outcome: Number of Participants With Improvement in Clinical Global Impression-Improvement (CGI-I) at 6 Weeks
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 121 | 57
Participants | 67 | 20
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change From Baseline in Pediatric Daytime Sleepiness Scale (PDSS) Scores at 6 Weeks
Description: The Pediatric Daytime Sleepiness Scale (PDSS) is an 8 question questionnaire scored on a scale from 0 (never) to 4 (always). Total scores range from 0 to 32, with increasing score reflecting greater sleepiness.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 121 | 57
Units on a Scale | -1.3 (5.36) | 0.9 (5.31)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.02, ANCOVA

8. Secondary Outcome: Change From Baseline in Pictorial Sleepiness Scale (PSS) Scores at 6 Weeks
Description: The Pictorial Sleepiness Scale (PSS) scores range from 1 (far left wide awake face) to 5 (far right very sleepy face). Increasing score reflects greater sleepiness.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 121 | 57
Units on a Scale | 0.0 (0.61) | 0.1 (0.63)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.231, ANCOVA

ADVERSE EVENTS:
Arm/Group | SPD503 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/121 | 0/57
Other Adverse Events (participants affected / at risk) | 96/121 | 32/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 (N=121) | Placebo (N=57)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Moderate loss of consciousness (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 (N=121) | Placebo (N=57)
Ear pain (Ear and labyrinth disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 10 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1
Fatigue (General disorders) | 6 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 0
Headache (Nervous system disorders) | 30 | 11
Sedation (Nervous system disorders) | 9 | 3
Somnolence (Nervous system disorders) | 50 | 13
Insomnia (Psychiatric disorders) | 3 | 1
Irritability (Psychiatric disorders) | 6 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.